CLINICAL TRIAL: NCT06221969
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) 2.4 mg/2.4 mg s.c. Once Weekly Versus Tirzepatide 15 mg s.c. Once Weekly in Participants With Type 2 Diabetes Inadequately Controlled on Metformin With or Without an SGLT2 Inhibitor
Brief Title: A Research Study to See How Much CagriSema Lowers Blood Sugar and Body Weight Compared to Tirzepatide in People With Type 2 Diabetes Treated With Metformin With or Without an SGLT2 Inhibitor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9388-4894; U1111-1282-5561 (Other: World Health Organization (WHO)); 2023-503789-21-00 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive cagrilintide dose 1 and semaglutide dose 2 subcutaneously once-weekly (dose escalation period of 16 weeks) for up to 68 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Tirzepatide (Active Comparator): Participants will receive tirzepatide dose 1 subcutaneously once-weekly (dose escalation period of 20 weeks) for up to 68 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously.
  Arms: CagriSema
Drug: Semaglutide — Semaglutide will be administered subcutaneously.
  Arms: CagriSema
Drug: Tirzepatide — Tirzepatide will be administered subcutaneously.
  Arms: Tirzepatide

SUMMARY:
This study will look at how well CagriSema helps people with type 2 diabetes lower their blood sugar and body weight. CagriSema is a new investigational medicine. Doctors may not yet prescribe CagriSema. CagriSema will be compared to a medicine called tirzepatide that doctors may prescribe in some countries. Participants will get either CagriSema or tirzepatide. Which treatment participant get is decided by chance like flipping a coin. Participant will have an equal chance of receiving either drug. For each participant, the study will last for up to one and a half years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes ≥ 180 days before screening.
* Stable daily dose(s) ≥ 90 days before screening of any of the following antidiabetic drug(s) or combination regimen(s) at effective or maximum tolerated dose as judged by the investigator: metformin with or without an sodium-glucose co-transporter-2 (SGLT2) inhibitor.
* HbA1c 7.0-10.5% (53-91 mmol/mol) (both inclusive) as determined by central laboratory at screening.
* Body mass index (BMI) of ≥ 30.0 kilogram per square meter (kg/m^2) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Renal impairment with estimated Glomerular Filtration Rate < 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) as determined by central laboratory at screening.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)-points.
Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%).

SECONDARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to end of treatment (week 68)
  Measured in %-points.
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimoles per liter (mmol/L).
Achievement of HbA1c target values of less than (<) 7.0% (<53 millimole per mole [mmol/mol]) | At end of treatment (week 68)
  Count of participant
Achievement of HbA1c target values of less than or equal to (≤) 6.5% (≤ 48 mmol/mol) | From baseline (week 0) to end of treatment (week 68)
  Count of participant
Achievement of greater than or equal to (≥) 5% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant
Achievement of ≥ 10% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant
Achievement of ≥ 15 % weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant
Achievement of ≥ 20 % weight reduction | From baseline (week 0) to end of treatment (week 68)
  Count of participant
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeters of mercury(mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 68)
  Measured in mmHg.
Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeter (cm).
Ratio to baseline in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: non-HDL cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Change From Baseline in Short Form-36 Version 2 (SF-36v2) (Acute Version) Health Survey | From baseline (week 0) to end of treatment (week 68)
  The SF-36 v2 will be used to measure differences in quality of life and mental wellbeing. The scores 0-100 (where higher scores indicated a better quality of life and mental wellbeing) from the SF-36 will be converted to a norm-based score using a T-score transformation in order to obtain a direct interpretation in relation to the distribution of the scores in the 1998 United States general population. Measured as score on a scale.
Change in Impact of Weight on Quality of Life-Lite Clinical Trials (IWQOL-Lite-CT) version 3 | From baseline (week 0) to end of treatment (week 68)
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Composite scores (score range): Physical composite (0-100), Psychosocial composite (0-100), Physical Function composite (0-100). Total score (0-100). Higher scores indicate better level of functioning.
Number of Treatment-emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 74)
  Count of events
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (<54 milligram per deciliter [mg/dL]), confirmed by blood glucose meter) | From baseline (week 0) to end of study (week 74)
  Count of episodes
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to end of study (week 74)
  Count of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (194):
- United States (116):
  - Synexus Clin Res-Birmingham, Birmingham, Alabama
  - Univ of Alabama_Birmingham, Birmingham, Alabama
  - Prime Medical Group, LLC, Gilbert, Arizona
  - Velocity Clinical Research-Phoenix, Phoenix, Arizona
  - Synexus Rsch /Cnt Phnx Med C, Phoenix, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Unity Health-Searcy Medical Center, Searcy, Arkansas
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - Headlands Research California, LLC, Escondido, California
  - Neighborhood Healthcare, Escondido, California
  - St. Jude Heritage Yorba Linda - Pediatric Ste D, Fullerton, California
  - Diabetes & Endocrine Specialists - La Mesa, La Mesa, California
  - Diabetes and Endocrine Specialists - La Mesa, La Mesa, California
  - Velocity Clin Res San Diego, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - Loma Linda Univ Hlth Cr Endo, Loma Linda, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Healthcare, Palm Springs, California
  - Velocity Clin Res - Panorama, Panorama City, California
  - Western University of Health Sciences, Pomona, California
  - Endocrinology Josel Cabaccan, San Jose, California
  - Mills-Peninsula Medical Center, San Mateo, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Premier Medical Center, Inc., Toluca Lake, California
  - Velocity Clin Res - Panorama, Van Nuys, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Optumcare Clinical Trials,LLC-Golden, Colorado Springs, Colorado
  - Northeast Res Inst. Inc., Jacksonville, Florida
  - Clinical Trial Services Corp, Miami, Florida
  - Bioclinical Research Alliance, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - South Broward Research LLC, Miramar, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Optimal Research Sites, Orange City, Florida
  - Trans Res Inst for Met & Diab, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - Center for Adv Res & Education, Gainesville, Georgia
  - Urban Family Practice Assoc, Marietta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Pacific Diabetes & Endo Ctr, Honolulu, Hawaii
  - St. Luke's Health System, Boise, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Clinical Invest Special_Gurnee, Gurnee, Illinois
  - Endeavor Health, Skokie, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - American Health Network of Indiana, LLC_Greenfield, Greenfield, Indiana
  - Iowa Diabetes & Endo Res Ctr, West Des Moines, Iowa
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - Velocity Clin Res Lafayette, Lafayette, Louisiana
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - International Diabetes Center, Minneapolis, Minnesota
  - Belzoni Clinical Research, Belzoni, Mississippi
  - Velocity Clin Res Gulfport, Gulfport, Mississippi
  - Diabetes & Endo Specialists Inc, Chesterfield, Missouri
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - Velocity Clin Res Albuquerque, Albuquerque, New Mexico
  - AMC Community Endocrinology, Albany, New York
  - Velocity Clin Res Syracuse, East Syracuse, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - UNC Eastowne Clinical Research Unit, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lucas Research Inc., Morehead City, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Remington Davis Inc, Columbus, Ohio
  - Advanced Medical Research, Maumee, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - CCT Research, Horsham, Pennsylvania
  - Thomas Jefferson University_Philadelphia, Philadelphia, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Velocity Clin Res Providence, East Greenwich, Rhode Island
  - Velocity Clinical Res-Anderson, Anderson, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Holston Medical Group Pc, Bristol, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - HealthStar Physicians PC, Morristown, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Velocity Clin Res, Austin, Texas
  - UT Health University of Texas, Bellaire, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Synexus Clin Res Dallas, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - JCCT- Juno NW Houston, Houston, Texas
  - Discovery MM Services, Inc, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Fmc Science, Llc, Lampasas, Texas
  - Quality Clinical Research, Inc., San Antonio, Texas
  - University of Texas San Antonio, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Mt Olympus Medical Research, LLC, Sugar Land, Texas
  - DM Clin Rsrch/Fam Diag Clinic, Tomball, Texas
  - Foothill Family Clinic South, Salt Lake City, Utah
  - J.Lewis Research Inc, South Jordan, Utah
  - Velocity Clin Res-Salt Lk City, West Jordan, Utah
  - TPMG Clinical Research, Newport News, Virginia
  - Rainier Clin Res Ctr Inc, Renton, Washington
  - Prevea Health, Green Bay, Wisconsin
- Argentina (10):
  - Buenos Aires Mácula, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CICEMO- Consultorio de Investigación Clínica EMO, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Medico Especializado_Capital Federal, Ciudad de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Metabolicas (IDIM), Buenos Aires
  - OMI- Organización Médica de Investigación, Buenos Aires
  - CICEMO- Consultorio de Investigación Clínica EMO, Buenos Aires
  - CEDIC Centro de Investigación Clínica, CABA
  - Centro de Investigación Clínica, CABA
  - Instituto de Investigaciones Clinicas Mar Del Plata, Mar del Plata
  - CEDIR - Centro de diagnóstico y rehabilitación Santa Fe, Santa Fe
- Australia (11):
  - Paratus Clinical, Blacktown, New South Wales
  - Paratus Clinical, Kanwal, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - University of Sunshine Coast, Morayfield, Queensland
  - Momentum Clinical Research, Taringa, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Austrials, St Albans, Victoria
  - Momentum Clinical Research, St Albans, Victoria
- Canada (19):
  - Centricity Research Calgary Endocrinology, Calgary, Alberta
  - Guilford Med Clinic, Surrey, British Columbia
  - TLC Diabetes and Endocrinology, Surrey, British Columbia
  - Ocean West Research Clinic, Surrey, British Columbia
  - Hilltop Medical Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Milestone Research, London, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Centre Medical Acadie, Montreal, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Centricity Research Oshawa, Barrie, West Oshawa
  - Clin des Mal Lipid de Quebec, Québec
  - Centre de Recherche Saint-Louis, Québec
- Colombia (5):
  - Clinica de la Costa, Barranquilla, Atlántico
  - FOSCAL, Floridablanca, Santander Department
  - Cimedical, Barranquilla
  - UNIENDO, Bogotá
  - Centro de Investigación en Reumatología y Especialidades Médicas S.A.S. CIREEM S.A.S., Bogotá
- India (20):
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - SSG Hospital, Baroda, Vadodara, Gujarat
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Indian Institute of Diabetes, Thiruvnanthapuram, Kerala
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - BSES MG hospital, Mumbai, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Maulana Azad Medical College, Delhi, New Delhi
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - AIG Hospitals,Hyderabad, Hyderabad, Telangana
  - Government Institute of Medical Sciences, Noida, Uttar Pradesh
  - BP Poddar Hospital, Kolkata, West Bengal
  - Rajiv Gandhi Centre for Diabetes and Endocrinology, J.N Medical College, Aligarh Muslim University, Aligarh
  - SRM Centre for Clinical Trials & Research, Chennai
  - Nirmal Hospital Pvt. Ltd., Surat
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram
- South Africa (6):
  - Dr Wilhase's rooms, Boksburg, Gauteng
  - Ubuntu Clinical Research, Johannesburg, Gauteng
  - Krugersdorp Medical Centre, Krugersdorp, Gauteng
  - Synapta Clinical Research Centre, Durban, KwaZulu-Natal
  - Dr J Reddy, Durban, KwaZulu-Natal
  - Bella Vita Clinical Research, Cape Town, Western Cape
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com